CLINICAL TRIAL: NCT01624519
Title: Agreement Between Arterial, Central Venous, and Peripheral Venous Lactate in the Intensive Care Unit
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of California, Los Angeles (Other)
Collaborators: Olive View-UCLA Education & Research Institute (Other)
Responsible Party: Principal Investigator, Richard Treger, Principal Investigator, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 10H-821002
Record Dates: First submitted 2012-06-18; First posted 2012-06-20 (Estimated); Last update posted 2012-06-20 (Estimated); Status verified 2012-06

CONDITIONS: Blood Lactate Analysis
Keywords: Arterial Lactate; Central Venous Lactate; Peripheral Venous Lactate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Other)
  Interventions: Procedure: Blood Lactate Analysis

INTERVENTIONS:
Procedure: Blood Lactate Analysis — When an arterial lactate is deemed to be necessary as part of ICU management, a central venous and peripheral venous sample will also obtained within 5 minutes. All of the samples will be analyzed using the same analyzer as quickly as possible.

SUMMARY:
The main objective of this study is to examine the agreement between arterial, central venous, and peripheral venous lactate values in a population of medical Intensive Care Unit (ICU) patients.

DETAILED DESCRIPTION:
This study is a single-center, prospective trial to assess the agreement between arterial, central venous, and peripheral venous lactate measurements. When an arterial lactate is deemed to be necessary as part of ICU management, a central venous and peripheral venous sample will also obtained within 5 minutes. All of the samples will be analyzed using the same analyzer as quickly as possible. A maximum of 10 paired arterial and venous lactate samples will be obtained per patient to prevent a single patient from dominating the data set. Additional data collected on a standardized data collection form will include primary diagnosis, intubation status, use of inotropic agents, hypotension (defined as a systolic blood pressure < 90 mm Hg), ICU length of stay and mortality. The Bland-Altman method will be used to assess agreement between arterial (A), central venous(CV), and peripheral venous (PV) lactate measurements. Approximately 50 patients will be enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients 18 years or older
* Admitted to the Intensive Care Unit (ICU)
* Determined by their treating clinicians to require both a central venous line and arterial line

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2012-08; Primary Completion 2013-08 (Estimated); Study Completion 2013-08 (Estimated)

PRIMARY OUTCOMES:
Agreement between peripheral venous, central venous, and arterial lactate values in a population of medical Intensive Care Unit (ICU) patients. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Rick Treger, Principal Investigator — Olive View-UCLA

REFERENCES:
- [Background] BRODER G, WEIL MH. EXCESS LACTATE: AN INDEX OF REVERSIBILITY OF SHOCK IN HUMAN PATIENTS. Science. 1964 Mar 27;143(3613):1457-9. doi: 10.1126/science.143.3613.1457. PMID 14107454
- [Background] Cowan BN, Burns HJ, Boyle P, Ledingham IM. The relative prognostic value of lactate and haemodynamic measurements in early shock. Anaesthesia. 1984 Aug;39(8):750-5. doi: 10.1111/j.1365-2044.1984.tb06516.x. PMID 6476309
- [Background] Mizock BA. Controversies in lactic acidosis. Implications in critically ill patients. JAMA. 1987 Jul 24-31;258(4):497-501. doi: 10.1001/jama.1987.03400040095029. PMID 3599345
- [Background] Domino EF, Bartolini A, Kawamura H. Effects of reticular stimulation, d-amphetamine and scopolamine on acetylcholine release from the hippocampus of brainstem transected cats. Arch Int Pharmacodyn Ther. 1977 Feb;225(2):294-302. PMID 849076
- [Background] Rivers E, Nguyen B, Havstad S, Ressler J, Muzzin A, Knoblich B, Peterson E, Tomlanovich M; Early Goal-Directed Therapy Collaborative Group. Early goal-directed therapy in the treatment of severe sepsis and septic shock. N Engl J Med. 2001 Nov 8;345(19):1368-77. doi: 10.1056/NEJMoa010307. PMID 11794169
- [Background] Mortensen JD. Clinical sequelae from arterial needle puncture, cannulation, and incision. Circulation. 1967 Jun;35(6):1118-23. doi: 10.1161/01.cir.35.6.1118. No abstract available. PMID 6026202
- [Background] Criscuolo C, Nepper G, Buchalter S. Reflex sympathetic dystrophy following arterial blood gas sampling in the intensive care setting. Chest. 1995 Aug;108(2):578-80. doi: 10.1378/chest.108.2.578. PMID 7634906
- [Background] Weil MH, Michaels S, Rackow EC. Comparison of blood lactate concentrations in central venous, pulmonary artery, and arterial blood. Crit Care Med. 1987 May;15(5):489-90. PMID 3568712
- [Background] Murdoch IA, Turner C, Dalton RN. Arterial or mixed venous lactate measurement in critically ill children. Is there a difference? Acta Paediatr. 1994 Apr;83(4):412-3. doi: 10.1111/j.1651-2227.1994.tb18131.x. PMID 8025400
- [Background] Middleton P, Kelly AM, Brown J, Robertson M. Agreement between arterial and central venous values for pH, bicarbonate, base excess, and lactate. Emerg Med J. 2006 Aug;23(8):622-4. doi: 10.1136/emj.2006.035915. PMID 16858095
- [Background] Gallagher EJ, Rodriguez K, Touger M. Agreement between peripheral venous and arterial lactate levels. Ann Emerg Med. 1997 Apr;29(4):479-83. PMID 9095008
- [Background] Younger JG, Falk JL, Rothrock SG. Relationship between arterial and peripheral venous lactate levels. Acad Emerg Med. 1996 Jul;3(7):730-4. doi: 10.1111/j.1553-2712.1996.tb03502.x. No abstract available. PMID 8816193
- [Background] Adams J 2nd, Hazard P. Comparison of blood lactate concentrations in arterial and peripheral venous blood. Crit Care Med. 1988 Sep;16(9):913-4. doi: 10.1097/00003246-198809000-00021. No abstract available. PMID 3402237
- [Background] Klein WW, Brandt D, Kraft-Kinz J, Schreyer H. [Dynamics and metabolism in coronary heart disease before and after revascularization intervention]. Acta Med Austriaca. 1976;3(3):69-73. German. PMID 1087300